CLINICAL TRIAL: NCT04369755
Title: Pilote Study : Brain Exploration in Magnetic Resonance Imaging in Parallel Transmission Mode (pTX) at 7 Tesla on Healthy Subject at Poitiers University Hospital
Brief Title: MR7T-Healthy-PTX : Brain Exploration in Magnetic Resonance Imaging in Parallel Transmission Mode (pTX) at 7 Tesla
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-A02689-48
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: MRI; PTX; BRAIN; 7 TESLA
Keywords: MRI; PTX; BRAIN; 7 TESLA

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI (Other): A MRI on PTX mode will be done on healthy subjects (approx. 90 min of sequences)
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — A MRI in PTX mode will be done on healthy subject (approx. 90 min of sequences)

SUMMARY:
Magnetic resonance imaging (MRI) is a non-invasive imaging modality used in routine clinical practice for clinical diagnosis by visualizing the anatomical structure and in vivo function of certain organs. The development of ultra-high field MRI systems with 7.0-T or higher, gives access to a new field of exploration of the human body by improving the speed of acquisition but also a better signal-to-noise ratio (SNR) and better resolution. In order to fully exploit the potential of these ultra-high field MRI scanners, various technical issues must be adressed. Indeed, the non-uniformity of the transmission field is one of them leading to non-uniform images with spatially varying contrast. Thus the pTX (parallel transmission) mode using multiple transmission channels allows spatial and temporal control over the RF waves.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Subject with no MRI contraindications (metallic shine, pacemaker)
* Free subject, without guardianship or curatorship or subordination
* A person affiliated to or beneficiary of a social security scheme.
* Informed and signed consent by the healthy volunteer after clear and fair information about the study

Exclusion Criteria:

* Subject with a contraindication to MRI (pregnancy, ocular metallic foreign body (accidental or other shrapnel); pacemaker (cardiac stimulator), implantable defibrillator, non MRI 7.0 T compatible neurostimulator, cochlear implants and generally any irremovably implanted electronic medical device; metallic heart valve, vascular clips formerly implanted on cranial aneurysm), metallic prostheses.
* Healthy volunteers suffering from claustrophobia
* Persons not benefiting from a Social Security scheme or not benefiting from it through a third party.
* Persons benefiting from reinforced protection, i.e. minors, pregnant and breastfeeding women, persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social institution, adults under legal protection and finally, patients in emergency situations.
* Pregnant or breastfeeding women, women of childbearing age who do not have effective contraception (hormonal/mechanical: per os, injectable, transcutaneous, implantable, intrauterine device, or surgical: tubal ligation, hysterectomy, total oophorectomy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-06-25 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the improvement of the Signal to Noise Ratio (SNR) in parallel transmission mode (pTx) versus without pTx at 7.0 T on different cerebral anatomical regions/structures (central gray nuclei, cerebellum, white matter, cortex). | 1 year
  The main evaluation criterion is the value of the signal-to-noise ratio in a global way but also by a unit comparison approach (voxel to voxel).
  It will be a question of linking these variations to the flip angles but also to the probable inhomogeneities of the B1+ field.

SECONDARY OUTCOMES:
Evaluation of the body temperature | 1 year
  Measurement of body temperature in healthy volunteers using a forehead thermometer before and after examination
Evaluation of anxiety before, during and after the MRI | 1 year
  Measurement of the healthy subject's feelings about the exam (anxiety, heat, nausea) using a grid proposed at the end of the exam.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Poitiers, Poitiers, France